CLINICAL TRIAL: NCT02910973
Title: Using a Transcutaneous Electrical Auricular Stimulator to Harness the Cholinergic Anti-Inflammatory Pathway
Acronym: TEACAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, Cynthia Aranow, MD, Investigator, Northwell Health
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: HS16-0530
Record Dates: First submitted 2016-09-20; First posted 2016-09-22 (Estimated); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Healthy Volunteers
Keywords: Inflammation, Vagus Nerve Stimulation
MeSH Terms: conditions — Inflammation | interventions — Vagus Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vagus Nerve Stimulation (Active Comparator): Device: Vagus nerve stimulation Patients will receive transcutaneous stimulation of the auricular branch of the left vagus nerve for 5 minutes.
  Interventions: Device: Vagus Nerve Stimulation
- Sham Vagus Nerve Stimulation (Sham Comparator): Patients will receive sham transcutaneous stimulation of the auricular branch of the left vagus nerve for 5 minutes.
  Interventions: Device: Sham Vagus Nerve Stimulation

INTERVENTIONS:
Device: Vagus Nerve Stimulation — Patients will receive transcutaneous stimulation of the auricular branch of the left vagus nerve for 5 minutes. Blood will be withdrawn prior to stimulation and 1 hour following the stimulation. The device is a handheld electrical pulse generator and a pair of electrodes to be placed at the ear for stimulation. The specific target at the ear will be the auricular branch of the vagus nerve which innervates the skin of the ear canal. Electrodes will be placed near/at the entrance to the canal of the ear to provide stimulation to the auricular branch of the vagus nerve.
  Arms: Vagus Nerve Stimulation
Device: Sham Vagus Nerve Stimulation — Patients will receive sham transcutaneous stimulation of the auricular branch of the left vagus nerve for 5 minutes. Blood will be withdrawn prior to stimulation and 1 hour following the stimulation. Sham stimulation will be performed in the identical manner as true transcutaneous stimulation except that the patient will not receive electrical stimulation of the vagus nerve.
  Arms: Sham Vagus Nerve Stimulation

SUMMARY:
Persistent chronic inflammation is an important underlying event in multiple diseases including rheumatoid arthritis, inflammatory bowel diseases and type 2 diabetes. These disorders are characterized as inflammatory in part because of the important mediating role of pro-inflammatory cytokines in their pathogenesis. This study will investigate whether transcutaneous auricular electrical stimulation of the vagus nerve will affect and decrease the inflammatory cytokine response in healthy individuals.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18-60 years,
2. Currently healthy with no medical problems
3. Able and willing to give written informed consent and comply with the requirements of the study protocol.

Exclusion Criteria:

1. History of any of the following: cardiac arrhythmia, coronary artery disease, autoimmune disease, chronic inflammatory disease, anemia, malignancy, depression, neurologic disease, diabetes mellitus, renal disease, malignancy, dementia, psychiatric illness including active psychosis, or any other chronic medical condition.
2. Family history of inflammatory disease
3. Treatment with an anti-cholinergic medication, including over the counter medications,
4. Implantable electronic devices such as pacemakers, defibrillators, hearing aids, cochlear implants or deep brain stimulators.
5. Current tobacco or nicotine user (to limit potential confounding effects of exposure to nicotine),
6. Chronic inflammatory disorders
7. Investigational drug and/or treatment during the 28 days or seven half-lives of the investigational drug prior to the start of study drug dosing (Day 0), whichever is the greater length of time,
8. Any condition which, in the opinion of the investigator, would jeopardize the subject's safety following exposure to a study intervention,
9. Pregnancy or lactation (Pregnancy status & lactation will be determined via self-report),
10. Implanted vagus nerve stimulator
11. Inability to comply with study procedures
12. Ear infection (otitis media or externa)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2023-12-13 (Actual); Study Completion 2023-12-13 (Actual)

PRIMARY OUTCOMES:
Lipopolysaccharide stimulated levels of TNF in whole blood. | 4 hours
  Whole blood will be taken from patients and stimulated by lipopolysaccharide. Levels of TNF produced by the cells in the whole blood after 4 hours of incubation will be measured.

SECONDARY OUTCOMES:
Lipopolysaccharide stimulated levels of cytokines such as IL-1, IL-6, IL-8, IL-10 and HMGB1 in whole blood. | 4 hours
  Whole blood will be taken from patients and stimulated by lipopolysaccharide. Levels of cytokines such as IL-1, IL-6, IL-8, IL-10 and HMGB1 that are produced by the cells in the whole blood after 4 hours of incubation will be measured.
Percentage of subjects with treatment emergent adverse events | 1 hour
  The percentage of participants with treatment emergent adverse events will be assessed using the NCI-CTAEversion4.

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Aranow, MD, Principal Investigator — Northwell Health
Locations (1):
- Feinstein Institute, Manhasset, New York, United States

IPD SHARING:
Plan to Share IPD: No